CLINICAL TRIAL: NCT03075488
Title: Ultrasound Pre-procedural Scan vs Conventional Landmark-guided Technique in Spinal Anesthesia in Orthopedic Obese Patients
Brief Title: Ultrasound Prescan vs Conventional Landmark-guided Technique in Spinal Anesthesia in Orthopedic Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Daniela Ghisi, principal investigator, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IOR-ACCURO
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2018-07

CONDITIONS: Ultrasonography; Anesthesia, Spinal; Body Mass Index; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional landmark-guided technique (Active Comparator): In this arm spinal anesthesia will be performed by using conventional cutaneous landmarks
  Interventions: Procedure: cutaneous landmarks
- Accuro device guided technique (Experimental): In this arm spinal anesthesia will be performed only after having detected the intralaminar space, the mid-line, the depth and the orientation for spinal needle insertion with pre-procedural scan performed with Accuro device
  Interventions: Device: Accuro

INTERVENTIONS:
Device: Accuro — spinal anesthesia injection based on identification of entry site with pre-procedural ultrasound scan with Accuro device
  Arms: Accuro device guided technique
Procedure: cutaneous landmarks — spinal anesthesia injection based on identification of entry site with palpation of cutaneous landmarks
  Arms: Conventional landmark-guided technique

SUMMARY:
The study is aimed at evaluating whether ultrasound pre-procedural scan with Accuro may reduce needle redirections when performing spinal injection in patients with BMI = or > 30 in orthopedic surgery

DETAILED DESCRIPTION:
This is a open-label randomised controlled study.

90 patients will be recruited and divided into two groups of 45 patients per group.

Patient recruitment will be performed by patient visit and checking inclusions and exclusion criteria. After written informed consent, every single patient will be allocated in one of the two groups following a computer generated randomization list.

Patients in both groups will undergo:

* standard monitoring with Non Invasive Blood Pressure (NIBP) cuff, three-lead electrocardiography (ECG) and Pulse-oximetry (SpO2).
* Peripheral intravenous access
* Sedation (as prescribed by the OR anesthesiologist)
* Spinal anesthesia performed by anesthesiologists skilled in both techniques (conventional landmark technique or Accuro guided) at the L3-L4, L4-L5 or L5-S1 level, with a 25 or 27 Gauge needle, with the surgical side declive or proclive according to the baricity of the local anesthetic used (sitting position, when needed, will be reported in the CRF)

In both groups an observer will monitor and register spinal procedure duration (starting point: anesthesiologist wearing sterile gloves, ending point: end of local anesthetic injection).

Control group (landmark technique):

The anesthesiologist will identify lumbar spinous processes with traditional landmark palpation. Once the correct interspinous level and the mid-line will be identified, the anesthesiologist will proceed with needle insertion and spinal injection.

Treatment group (ultrasound pre-procedural scan with Accuro):

By using Accuro US probe the anesthesiologist will perform a pre-procedural lumbar spine scan to detect the needle entry site. After image optimization, the Accuro probe will be aligned with the spine mid-line, as indicated by a dashed red-line on the screen. After that the interlaminar space at the desired intervertebral level will be detected, as indicated by orange overlay in the screen. The depth and the device angle used to detect the interlaminar space will be annotated. The anesthesiologist will then disengage the Accuro Locator needle guide and press gently against the skin. Then the probe will be removed and the spinal injection will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* BMI ≥ 30 kg/m2
* American Society of Anesthesiologists' (ASA) classification I-III
* Orthopedic surgery to be performed under spinal anesthesia
* Able to understand and to sign informed consent

Exclusion Criteria:

* Local anaesthetic allergy
* Serious spine deformities
* Previous spine surgery
* Inability to express informed consent
* Contraindications to spinal anaesthesia
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Needle redirections | duration of spinal injection procedure
  To evaluate if there is a significant difference about numbers of needle redirections between conventional landmark guided technique and Accuro device guided technique

SECONDARY OUTCOMES:
Number of needle insertions | duration of spinal injection procedure
  Number of needle insertions through the skin
Procedure duration | duration of spinal injection procedure
  Procedure duration from steril gloves wearing to the end of the spinal anesthetic injection
Side effects and complications | 36 months
  To check if present side effects and complications during the procedure
Procedure failure | duration of surgical procedure
  To check eventually procedure failure and the need of using alternative anesthesia technique
Patient satisfaction | 24 hours
  Evaluation of patient satisfaction and procedure-related pain 24 hours after spinal injection

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghisi D, Tomasi M, Giannone S, Luppi A, Aurini L, Toccaceli L, Benazzo A, Bonarelli S. A randomized comparison between Accuro and palpation-guided spinal anesthesia for obese patients undergoing orthopedic surgery. Reg Anesth Pain Med. 2019 Oct 25:rapm-2019-100538. doi: 10.1136/rapm-2019-100538. Online ahead of print. PMID 31653795